CLINICAL TRIAL: NCT05113342
Title: Phase I/IIa Study of Descartes-25 in Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: Descartes-25 in Relapsed/Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Phase 1 enrollment completed. Further clinical development terminated.
Sponsor: Cartesian Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DC25-1A
Record Dates: First submitted 2021-10-19; First posted 2021-11-09 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Multiple Myeloma; Relapse Multiple Myeloma
Keywords: myeloma; multiple myeloma; Relapse Refactory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm 1: Dose Level 1 (Experimental): Minimum of 3 patients per Dose Level will be treated sequentially with once weekly infusions for 3 weeks in a 28-day cycle until the Maximum Tolerated Dose (MTD) is reached.
  Interventions: Drug: Descartes-25
- Arm 2: Dose Level 2 (Experimental): Minimum of 3 patients per Dose Level will be treated sequentially with once weekly infusions for 3 weeks in a 28-day cycle until the Maximum Tolerated Dose (MTD) is reached.
  Interventions: Drug: Descartes-25
- Arm 3: Dose Level 3 (Experimental): Minimum of 3 patients per Dose Level will be treated sequentially with once weekly infusions for 3 weeks in a 28-day cycle until the Maximum Tolerated Dose (MTD) is reached.
  Interventions: Drug: Descartes-25
- Arm 4: Dose Expansion (Experimental): In Arm 2, the MTD established in Arm 1 will be administered for 3 28-day cycles to further evaluate the product's safety and preliminary efficacy.
  Interventions: Drug: Descartes-25

INTERVENTIONS:
Drug: Descartes-25 — allogeneic Mesenchymal Stem Cell product.
  Other Names: DC-25

SUMMARY:
This is a Phase I/IIa dose-escalation study to evaluate the safety, tolerability, and preliminary efficacy of an allogeneic Mesenchymal Stem Cell (Descartes-25) product secreting a bispecific protein and other proteins in patients with Relapsed/Refractory Multiple Myeloma.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older'
* diagnosed with active R/RMM, who have failed 2 lines of treatment
* have measurable disease

Exclusion Criteria:

- Patients with active plasma cell leukemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-11-25 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2024-11-08 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 1 Year
  Dose Level at which no more than 20% of the patients treated have shown Dose-Limiting Toxicity.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Louisiana State University Health Science Center at Shreveport, Shreveport, Louisiana
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
- Saglik Bilimleri Universitesi, Ankara, Anatolia, Turkey (Türkiye)